CLINICAL TRIAL: NCT03488433
Title: Randomized Controlled Trial Comparing Abduction Shoulder Brace Versus Antirotation Sling for Postoperative Immobilization Following Reverse Total Shoulder Arthroplasty and Rotator Cuff Repair
Brief Title: Abduction Brace Versus Antirotation Sling for Immobilization Following Reverse Shoulder Arthroplasty and Rotator Cuff Repair
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI institutional transition prior to enrollment
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, H Mike Kim, Associate Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00008723
Record Dates: First submitted 2017-12-21; First posted 2018-04-05 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Rotator Cuff Tear Arthropathy; Rotator Cuff Tear
Keywords: Postoperative shoulder immobilization; Reverse total shoulder arthroplasty; Neutral rotation shoulder brace; Antirotation sling
MeSH Terms: conditions — Rotator Cuff Tear Arthropathy; Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: Patients undergoing reverse total shoulder arthroplasty or rotator cuff repair will be randomly assigned to two groups of immobilization method groups, namely abduction brace group and antirotation sling group.
Masking Description: Patients will be randomly assigned to either neutral rotation brace, or antirotation sling following reverse total shoulder arthroplasty. The patients, PI and co-investigators all will be blinded to patient assignments until the day of surgery when an envelope with their assignments are given to surgeon at day of surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Antirotation sling (Active Comparator): Patients who undergo reverse shoulder arthroplasty or rotator cuff repair will be randomly assigned to this group.
  Interventions: Device: Antirotation sling
- abduction brace (Active Comparator): Patients who undergo reverse shoulder arthroplasty or rotator cuff repair will be randomly assigned to this group.
  Interventions: Device: Abduction brace

INTERVENTIONS:
Device: Abduction brace — Donjoy Ultrasling IV
  Arms: abduction brace
Device: Antirotation sling — Donjoy shoulder immobilizer
  Arms: Antirotation sling

SUMMARY:
To compare the functional and anatomical outcomes, and patient satisfaction and compliance between two different postoperative immobilization methods - abduction shoulder brace versus simple arm sling - following 2 common shoulder surgical procedures - rotator cuff repair (RCR) and reverse total shoulder arthroplasty (RTSA) through a prospective randomized clinical trial.

DETAILED DESCRIPTION:
Scientific Background and Gaps Rotator cuff repair and reverse total shoulder arthroplasty are common procedures that aim to provide patients with less pain, better shoulder function, and overall improved quality of life. The number of these procedures performed annually has increased dramatically, and improved outcomes have been demonstrated for each intervention. Part of the success of these operations is dependent on postoperative rehabilitation and patient compliance. Shoulder immobilization versus early range of motion following each procedure has conflicting data, and recent studies have shown that the method of shoulder immobilization may not influence clinical outcomes. Previous studies, both clinical and biomechanical, have demonstrated that arm position following RCR impacts tension and stress placed on the repair, but few have shown whether this translates to improved patient outcomes. Some surgeons prefer simple arm slings for the above-named procedures, while others opt for the abduction brace. Multiple studies have shown the optimal shoulder position that places the least amount of tension on the RCR, or soft tissue envelope following RTSA, however there is no consensus as to the optimal postoperative immobilization technique that significantly affects patient outcomes. An antirotation sling is significantly cheaper than an abduction shoulder brace, and our anecdotal experience is that patients experience more difficulties with an abduction shoulder brace than an antirotation sling. Our study aims to determine whether patient outcomes are significantly affected by immobilization with an abduction brace or simple arm sling. Our hypothesis is that antirotation slings are no better or worse than shoulder abduction braces in regards to shoulder range of motion, satisfaction and compliance with the immobilization method, and pain.

Study Rationale There is a lack of evidence regarding abduction braces versus simple arm slings for postoperative immobilization following rotator cuff repair and reverse total shoulder arthroplasty. A better understanding of outcomes between each device will allow for more options available to the patient and surgeon, as well as a potential for decreased cost to the patient as there is a substantial difference in cost between the two devices.

ELIGIBILITY:
Inclusion Criteria:

* patients 18 years and above
* male or female Rotator cuff tear patients - adults with a small or medium-sized (less than 3 cm in the anteroposterior dimension) full-thickness tear of supraspinatus and/or infraspinatus tendon, diagnosed with MRI or ultrasound, unresponsive to conservative therapy for >3 months

Reverse total shoulder arthroplasty patients - adults with rotator cuff arthropathy, glenohumeral joint arthritis with significant glenoid wear or retroversion requiring reverse arthroplasty or massive irreparable rotator cuff tear, functional deltoid, as demonstrated on x-rays, MRI, and physical exam. Failed conservative management for >3 months

Exclusion Criteria:

* younger than 18 years old
* chronic opiate use, fibromyalgia
* Rotator cuff repair patients - no previous rotator cuff repair surgery, no concomitant preoperative stiffness (definition: < 30 degree passive external rotation, < 100 degree passive forward elevation), no concomitant full-thickness subscapularis tear, no neurologic disorder affecting the ipsilateral upper extremity, no concomitant cervical pathology, partial thickness tear, large or massive tears (>3cm in the anteroposterior dimension), glenohumeral or rotator cuff arthropathy, history of rheumatoid arthritis.
* Reverse total shoulder arthroplasty patients -no concomitant preoperative stiffness (definition: < 30 degree passive external rotation, < 100 degree passive forward elevation), no concomitant neurologic disorder affecting the ipsilateral upper extremity, no concomitant cervical pathology.

arthroplasty for fracture, revision surgery, insufficient bone stock requiring hemiarthroplasty, deltoid dysfunction, history of rheumatoid arthritis.

* prisoners
* non English speaking or unable to understand consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Postoperative range of motion | Measured at 6 weeks, 12 weeks, 5 months, and 12 months following the index procedure.
  Both active and passive range of motion will be measured in forward elevation, external rotation at the side, internal rotation at extension, external rotation at abduction, and internal rotation at abduction by the examiners using a handheld goniometer. Multiple time points are for assessing the changes in motion.

SECONDARY OUTCOMES:
Visual analog scale (VAS) pain score | Measured at 6 weeks, 12 weeks, and 5 months, and 12 months after surgery
  Measures subjective pain; minimum 0, maximum 10 with 0 being a pain-free condition and 10 being the worst pain ever experienced
American Shoulder and Elbow Surgeons (ASES) score | Assessed at 5 and 12 months after surgery
  Measures patient's subjective shoulder function using a series of survey questions regarding subjective rating of range of motion, strength, use, and pain of the shoulder; minimum 0 to maximum 100 with 0 being the worst shoulder function and 100 being the best shoulder function
Patient compliance 5-point Likert-type scale | Assessed at 12 weeks after surgery
  Measure compliance with their assigned immobilization method measured using a 5-point Likert-type scale (Question: Did you wear the sling as instructed in the protocol? Not at all, occasionally, about a half of the time, for the most part, yes definitely)
Patient satisfaction 5-point Likert-type scale | Measured at 12 weeks
  Measures overall patient satisfaction with their immobilization method using a 5-point Likert-type scale (Question: Are you satisfied with the immobilization method using the sling you wore? Not at all, not much, so-so, pretty much, yes definitely)
Complications | Assessed at 12 months after surgery
  Such as shoulder dislocations, wound healing issue, pain development at areas other than the operated shoulder due to the immobilization, etc
QuickDASH (Disability of arm, shoulder, and hand) score system | Assessed at 5 and 12 months after surgery
  Measures the extent of subjective disability of upper extremity; consisted of survey questions regarding subjective pain and function of the upper extremity; Minimum 0, maximum 100 with 0 being no disability and 100 being most severe disability)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kiet TK, Feeley BT, Naimark M, Gajiu T, Hall SL, Chung TT, Ma CB. Outcomes after shoulder replacement: comparison between reverse and anatomic total shoulder arthroplasty. J Shoulder Elbow Surg. 2015 Feb;24(2):179-85. doi: 10.1016/j.jse.2014.06.039. Epub 2014 Sep 9. PMID 25213827
- [Background] Lambers Heerspink FO, van Raay JJ, Koorevaar RC, van Eerden PJ, Westerbeek RE, van 't Riet E, van den Akker-Scheek I, Diercks RL. Comparing surgical repair with conservative treatment for degenerative rotator cuff tears: a randomized controlled trial. J Shoulder Elbow Surg. 2015 Aug;24(8):1274-81. doi: 10.1016/j.jse.2015.05.040. PMID 26189808
- [Background] Hollman F, Wolterbeek N, Zijl JAC, van Egeraat SPM, Wessel RN. Abduction Brace Versus Antirotation Sling After Arthroscopic Cuff Repair: The Effects on Pain and Function. Arthroscopy. 2017 Sep;33(9):1618-1626. doi: 10.1016/j.arthro.2017.02.010. Epub 2017 Apr 17. PMID 28427872
- [Background] Zuckerman JD, Leblanc JM, Choueka J, Kummer F. The effect of arm position and capsular release on rotator cuff repair. A biomechanical study. J Bone Joint Surg Br. 1991 May;73(3):402-5. doi: 10.1302/0301-620X.73B3.1670437.
- [Background] Conti M, Garofalo R, Castagna A. Does a brace influence clinical outcomes after arthroscopic rotator cuff repair? Musculoskelet Surg. 2015 Sep;99 Suppl 1:S31-5. doi: 10.1007/s12306-015-0357-0. Epub 2015 May 10. PMID 25957544
- [Background] Jackson M, Tetreault P, Allard P, Begon M. Optimal shoulder immobilization postures following surgical repair of rotator cuff tears: a simulation analysis. J Shoulder Elbow Surg. 2013 Aug;22(8):1011-8. doi: 10.1016/j.jse.2012.10.042. Epub 2013 Jan 24. PMID 23352183
- [Background] Pedowitz RA, Yamaguchi K, Ahmad CS, Burks RT, Flatow EL, Green A, Iannotti JP, Miller BS, Tashjian RZ, Watters WC 3rd, Weber K, Turkelson CM, Wies JL, Anderson S, St Andre J, Boyer K, Raymond L, Sluka P, McGowan R; American Academy of Orthopaedic Surgeons. Optimizing the management of rotator cuff problems. J Am Acad Orthop Surg. 2011 Jun;19(6):368-79. doi: 10.5435/00124635-201106000-00007. PMID 21628648
- [Background] Hatakeyama Y, Itoi E, Pradhan RL, Urayama M, Sato K. Effect of arm elevation and rotation on the strain in the repaired rotator cuff tendon. A cadaveric study. Am J Sports Med. 2001 Nov-Dec;29(6):788-94. doi: 10.1177/03635465010290061901. PMID 11734494
- [Background] Mall NA, Tanaka MJ, Choi LS, Paletta GA Jr. Factors affecting rotator cuff healing. J Bone Joint Surg Am. 2014 May 7;96(9):778-88. doi: 10.2106/JBJS.M.00583. PMID 24806015